CLINICAL TRIAL: NCT01921569
Title: Micronized Dehydrated Human Amniotic Membrane (dHACM) Suspension in the Treatment of Lateral Epicondylitis.
Brief Title: Micronized Dehydrated Human Amniotic Membrane Suspension in the Treatment of Lateral Epicondylitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed by sponsor
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFLATEP001
Record Dates: First submitted 2013-07-18; First posted 2013-08-13 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Epicondylitis, Lateral Humeral
MeSH Terms: conditions — Tennis Elbow | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- dHACM (Experimental): Standard of Care Therapy plus dHACM injection at initial visit, to be repeated if symptoms persist at the time of week 4 and week 8 follow up visits.
  Interventions: Behavioral: Standard of Care Therapy; Other: dHACM Injection
- Saline Injection (Placebo Comparator): Standard of Care Therapy plus normal saline injection instead of active agent at initial visit, to be repeated if symptoms persist at the time of week 4 and week 8 follow up visits.
  Interventions: Behavioral: Standard of Care Therapy; Other: Normal Saline Injection

INTERVENTIONS:
Behavioral: Standard of Care Therapy — Rest, ice, compression, elevation (RICE), NSAID or salicylate medication for pain, Physical Therapy and stretching exercises, Reduction in impact activities, to include an arm sling.
Other: dHACM Injection — Injection into affected area with micronized dHACM suspended with total volume of 1 cc normal saline.
  Arms: dHACM
Other: Normal Saline Injection — Injection into affected area with 1.0 cc normal saline solution instead of active agent.
  Arms: Saline Injection

SUMMARY:
The purpose of this study is to determine whether micronized dehydrated human amniotic membrane (dHACM) suspension is more effective in reducing inflammation than conservative measures alone when used to treat acute/early lateral epicondylitis.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Medicare patients may be selected.
* Both male and female patients will be selected.
* A negative x-ray of the elbow
* Diagnosis of lateral epicondylitis by history and exam with symptoms for no longer than one year.
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
* Patient understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
* Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken.

Exclusion Criteria:

* Prior surgery at the site
* Site exhibits clinical signs and symptoms of infection.
* History of chronic soft tissue inflammation of more than 6 months.
* A positive X-ray for fracture or significant anatomic abnormality including fracture, advanced arthritis, excessive calcification, etc.
* No history of corticosteroid injection within the past 30 days.
* Joint instability
* No rheumatologic conditions involving the elbow.
* No evidence of significant neurological entrapment or neurological disease of the forearm
* Concurrent cervical radiculopathy
* The presence of comorbidities that can be confused with or can exacerbate the condition including:

  * Previous elbow trauma
  * Previous elbow surgery
* Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study. (i.e. a one month "washout period" for these drugs.)
* Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
* History of radiation at the site.
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
* Patients who are unable to understand the aims and objectives of the trial.
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment.
* Pregnant or breast feeding. No pregnancy within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving improvement in ASES elbow score in the dHACM treatment group vs the control group. | 12 weeks

SECONDARY OUTCOMES:
Proportion of patients achieving improvement in range of motion in the dHACM treatment group vs the control group. | 12 weeks

OTHER OUTCOMES:
Pain scores | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kremchek, MD, Principal Investigator — Beacon Orthopaedics & Sports Medicine
Locations (1):
- Beacon Orthopaedics & Sports Medicine, Sharonville, Ohio, United States